CLINICAL TRIAL: NCT05834777
Title: Prevention of Intradialytic Hypotension by Inhibiting Bradykinin B2 Receptor A Randomized, Double-blind, Placebo-controlled, Cross Over Explorative Study
Brief Title: Prevention of Intradialytic Hypotension by Inhibiting Bradykinin B2 Receptor
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Pharvaris Netherlands B.V. (Industry); Renal Research Institute (Other)
Responsible Party: Principal Investigator, Jorge Gamboa, Research Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 222301
Record Dates: First submitted 2023-02-27; First posted 2023-04-28 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Intradialytic Hypotension
Keywords: Hemodialysis; Intradialytic hypotension; Bradykinin; Kallikrein-Kinin System; Icatibant
MeSH Terms: interventions — icatibant

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, cross-over study, with a pharmocokinetics evaluation phase.
  Study duration for main cross-over study: Approximately 60 days including screening evaluation activities.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: For the procedure of the cross-over main study, both participating sites will recruit patients that will be randomized through a centralized randomization key to ensuring an equally balanced allocation of patients to the respective cross-over groups (icatibant or placebo). All study personnel will be blinded except the IDS pharmacy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Icatibant (Experimental): 153 mL 0.9% saline bag containing 30 mg icatibant acetate (10 mg/ml) IV at each dialysis treatment for four weeks (12 hemodialysis sessions)
  Interventions: Drug: Icatibant
- Placebo (Placebo Comparator): 153 mL 0.9% saline bag IV at each dialysis treatment at each dialysis treatment for four weeks (12 hemodialysis sessions)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Icatibant — Icatibant will be administered with an infusion rate of 100µg/kg/h for 15 minutes before their hemodialysis session (pre-infusion) and 50µg/kg/h during their routine hemodialysis session (maintenance infusion).
  Arms: Icatibant
Drug: Placebo — 0.9% sodium chloride will be administered as the same rate as icatibant
  Arms: Placebo

SUMMARY:
Currently, there is no medication available to adequately treat patients undergoing hemodialysis who are suffering from intradialytic hypotension (IDH). Medical interventions such as Trendelenburg positioning, saline bolus administration, reduction of ultrafiltration rate, interruption of the hemodialysis, and other medical treatments are the methods of choice to treat the hypotensive condition of these patients and thus to maintain the systolic blood pressure. Patients suffering from IDH have a higher reported mortality rate due to the given stress on their cardiovascular system. New treatments, therefore, would give clinicians an additional alternative to current existing approaches and might help patients to maintain their blood pressure during hemodialysis.

The main objective of the study is to evaluate the efficacy of icatibant in the prevention of systolic blood pressure (SBP) drop in patients on hemodialysis suffering from recurrent IDH episodes during hemodialysis.

DETAILED DESCRIPTION:
Aim 1 is to test the hypothesis that in patients prone to IDH, blockade of bradykinin B2 receptor with icatibant prevents the drop of blood pressure and maintains hemodynamic stability. For this purpose, heart rate and blood pressure during hemodialysis are monitored. Importantly, the study will be conducted in an outpatient clinic, using the patients' usual hemodialysis dose and settings as for a regular hemodialysis session.

Aim 2 is to test the hypothesis that in patients prone to IDH, inhibition of the plasma kallikrein system with icatibant prevents symptoms associated with IDH such as cramps, dizziness, and nausea, and improves the quality of life (QoL) and recovery time after hemodialysis. Hemodialysis is associated with many complications, including IDH, that negatively affect the QoL of patients and their families. Any intervention that prevents the occurrence of IDH will result in a faster recovery from hemodialysis. The present study will evaluate the impact of icatibant on preventing symptoms associated with IDH and reducing recovery time after hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 to ≤ 80 years of age
* Patients with end-stage renal disease on hemodialysis (including hemodiafiltration) for at least 6 months, receiving 3 dialysis sessions per week and who are in a stable clinical condition per investigator's judgement
* Patients on hemodialysis with at least 6 IDH episodes during the last 8 weeks based on medical record assessment
* Pre-dialysis systolic blood pressure ≥ 110 and ≤ 170 mmHg assessed by two consecutive and averaged pre-HD blood pressure measurments
* Patients adequately hemodialyzed with a Kt/V ≥ 1.2
* Patients whose treatment regimen remained unchanged within 14 days prior to dosing (diet, medication, dry weight, treatment time, dialysate composition and temperature, dialysis shift, blood flow, and dialysate flow, vascular access)
* Female subjects < 55 years of age to agree on effective contraception methods throughout the study period and who have a negative pregnancy test before initiating study activities
* Body weight ≤ 150 kg

Exclusion Criteria:

* Patients who have been hospitalized during the last 4 weeks before enrolment, except vascular access related hospitalization
* Patients with known clinically evident inflammatory or infectious disease per investigator's evaluation
* Severe anemia with a hemoglobin (Hb) < 8.0 g/dL at screening
* Platelet count < 50 x 109/L
* Hepatic disease associated with ALT > 3x ULN, or total bilirubin >2x ULN with direct bilirubin > 20% of the total bilirubin level
* Known bleeding disorders e.g., von-Willebrand disease or Hemophilia A, B, C, etc.
* Recent (<3 months before screening) thromboembolic event, e.g., acute coronary syndrome, stroke, or venous thrombosis embolism (except dialysis access thrombosis)
* Recent (<3 months before screening) major surgery or scheduled major surgery during study participation
* Scheduled living donor renal transplant during study participation
* Persistent heart failure as classified by the New York Heart Association (NYHA) classification of 3 or higher
* Receiving antiplatelet therapy except daily ASA ≤ 150 mg/day
* Receiving anticoagulation in therapeutic doses, other than standard anticoagulation during the hemodialysis procedure
* Patients with significant pre-dialysis overload as defined by > 5kg above dry weight estimated by bioimpedance spectroscopy
* Patient's life expectancy < 6 months per investigator's judgement

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Blood pressure during hemodialysis | 0-8 weeks
  Average systolic blood pressure

SECONDARY OUTCOMES:
Hypotension events | 0-8 week
  We will record the number of hypotensive events during hemodialysis. We expect a decrease of event in the treatment arm compared to placebo
Symptomatology associated with hypotension | 0-8 weeks
  At the end of each hemodialysis session in the cross-over main study, the presence of any symptoms associated with hypotension using a standardized questionnaire will be assessed. This questionnaire will include symptoms such as cramps, dizziness, nausea and fatigue rating, and will be scored according to the severity from 0 to 4 (none to severe) for the first listed symptoms, and according to the SONG-HD Fatigue scoring for the last listed symptom, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge L Gamboa, MD/PhD, Principal Investigator — Vanderbilt University Medical Center; Peter Kotanko, MD, FASN, Principal Investigator — Renal Research Institute; Talat A Ikizler, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt Fresenius, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No